CLINICAL TRIAL: NCT06080243
Title: A Phase II Randomised, Controlled Trial to Evaluate the Safety, Immunogenicity and Efficacy of the R21/Matrix-M1 Malaria Vaccine in Healthy African Women of Childbearing Potential in Mali
Brief Title: Assessment of Safety, Immunogenicity and Efficacy of R21/Matrix-M1 Malaria Vaccine in Healthy WOCBP in Mali
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: Malaria Research and Training Center, Bamako, Mali (Other); European Vaccine Initiative (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: VAC 094
Record Dates: First submitted 2023-08-28; First posted 2023-10-12 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Healthy Women of Child Bearing Potential
MeSH Terms: interventions — Sodium Chloride; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental-Standard Regime Malaria Vaccine Group1 (Active Comparator): Participants receiving three doses of R21/Matrix-M1 malaria vaccine at months 0, 1 and 2.
  Interventions: Biological: R21/Matrix-M1
- Experimental-Standard Regime Malaria Vaccine Group2 (Active Comparator): Participants receiving normal saline (placebo) at month 0 and two doses of R21/Matrix-M1 malaria vaccine at month 1 and 2
  Interventions: Biological: Saline and R21/Matrix-M1
- Experimental-Standard Regime Group3 (Active Comparator): Participants receiving three doses of normal saline (placebo) at months 0, 1 and 2
  Interventions: Other: Sterile isotonic (0.9%) normal saline

INTERVENTIONS:
Biological: R21/Matrix-M1 — 10 µg of R21 and 50 µg of Matrix-M1
  Arms: Experimental-Standard Regime Malaria Vaccine Group1
Biological: Saline and R21/Matrix-M1 — Saline and 10 µg of R21 and 50 µg of Matrix-M1
  Other Names: R21/Matrix-M1
  Arms: Experimental-Standard Regime Malaria Vaccine Group2
Other: Sterile isotonic (0.9%) normal saline — Saline
  Other Names: Placebo
  Arms: Experimental-Standard Regime Group3

SUMMARY:
This will be a double-blind, individually randomised trial, to assess the safety, tolerability, immunogenicity, and protective efficacy of two and three doses of the R21/Matrix-M1 malaria vaccine or placebo given at 4 week intervals in healthy women of childbearing potential (WOCBP), who are on pregnancy prevention during vaccination, but report plans to become pregnant in the near future.

Participants will be randomised in Year 1 into three groups in a 1:1:1 ratio:

* Arm 1 (n=110): will receive three doses of R21/Matrix-M1 malaria vaccine at months 0, 1 and 2.
* Arm 2 (n=110): will receive normal saline (placebo) at month 0 and two doses of R21/Matrix-M1 malaria vaccine at months 1 and 2.
* Arm 3 (n=110): will receive three of doses normal saline (placebo) at months 0, 1 and 2. In Year 2: Non-pregnant participants in arms 1 and 2 will be randomised in a 1:1 ratio to receive a booster dose of R21/Matrix-M1 malaria vaccine or placebo at the beginning of the malaria transmission season. Participants in the control group (arm 3) will receive normal saline (placebo).

Initial follow-up will be for two years after dose three, with an efficacy analysis at 6, 12, 18 and 24 months after dose 3.

Participants will be monitored for safety, tolerability, immunogenicity, and malaria infection during the follow-up period.

Participants will also be monitored for pregnancy over 12 months post primary and booster vaccination and those who become pregnant will be followed during their pregnancy and for 1 year post-delivery (as well as their offspring) for safety and malaria infection

DETAILED DESCRIPTION:
The design will be a double blind, placebo-controlled study. Malian adult WOCBP between 18 and 35 years of age who consent to participate will be randomised to receive R21/Matrix-M1vaccine or normal saline to assess the safety, immunogenicity and protective efficacy of R21/Matrix-M1 Vaccine.

Randomisation and Study Arms Consenting participants who have satisfied all the eligibility criteria and completed the baseline assessment will be individually randomised within the study groups using an electronic randomisation system into three arms in a 1:1:1 ratio.

* Arm 1: Participants will receive three doses of R21/Matrix-M1 malaria vaccine at months 0, 1 and 2.
* Arm 2: will receive normal saline (placebo) at month 0 and two doses of R21/Matrix-M1 malaria vaccine at month 1 and 2.
* Arm 3: will receive three doses of normal saline (placebo) at months 0, 1 and 2.

Participants will be assessed for safety, immunogenicity and efficacy for 12 months. After 12 months non-pregnant participants in arms 1 and 2, will be randomised in a 1:1 ratio; half in each of these two arms will receive a booster dose of R21/Matrix-M1 vaccine and half will receive a placebo injection (normal saline) and be followed up for an additional 12 months.

All injections will be administered intramuscularly in the deltoid region, preferably of the non-dominant arm. Post third injection, participants will be followed through the malaria transmission (rainy) season, approximately 6 months, and then the ensuing dry season for an additional 6 months. Participants will be monitored for safety, immunogenicity, and protective efficacy (malaria infection) during the follow-up period.

For any women who become pregnant during the two-year period (first year and second year) of the trial, follow up will continue through the end of pregnancy, and any viable newborns/infants and their mothers will be followed through the first year of life.

ELIGIBILITY:
Inclusion Criteria:

* Healthy females of childbearing potential aged ≥ 18 and ≤ 35 years
* Able and willing (in the Investigator's opinion) to comply with all study requirements.
* Agreement to release medical and other information concerning contra-indications for participation in the study, and to be attended by a study clinician for physical examination and any other clinical investigations.
* Provide written informed consent.
* Available for the duration of the study
* Must be willing to use reliable contraception (defined as: pharmacologic contraceptives [parental delivery] or pre-existing intrauterine or implantable device) from 21 days prior to study day 1 to 28 days after third vaccination and 21 days prior to the booster vaccination to 28 days after the booster vaccination.
* Report being interested in becoming pregnant within the next 1 year.

Exclusion Criteria:

* Pregnancy at the time of enrollment or any subsequent vaccination, as determined by a positive urine or serum human chorionic gonadotropin (β-hCG) test.
* Biologically unable to become pregnant secondary to: surgical sterilization, premature ovarian insufficiency (defined as no menses for ≥12 months without an alternative medical cause).
* Behavioral, cognitive, or psychiatric disease that in the opinion of the investigator affects the ability of the participant to understand and comply with the study protocol.
* Hemoglobin (Hgb), WBC, absolute neutrophils, and platelets outside the local laboratory-defined limits of normal and ≥ Grade 2 (participants may be included at the investigator's discretion for 'not clinically significant' abnormal values).
* Alanine transaminase (ALT) or creatinine (Cr) level above the local laboratory-defined upper limit of normal and ≥ Grade 2 (participants may be included at the investigator's discretion for 'not clinically significant' abnormal values).
* Infected with human immunodeficiency virus (HIV).
* Known or documented sickle cell disease by history or lab test at screening (Note: known sickle cell trait is NOT exclusionary).
* Evidence of clinically significant neurologic, cardiac, pulmonary, hepatic, endocrine, rheumatologic, autoimmune, hematological, oncologic, or renal disease by history, physical examination, and/or laboratory studies including urinalysis.
* Participation in another research study involving receipt of an investigational product in the 30 days preceding enrolment or during the trial follow up period.
* Medical, occupational, or family problems as a result of alcohol or illicit drug use during the past 12 months.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine.
* History of hereditary angioedema acquired angioedema, or idiopathic angioedema.
* History of a severe allergic reaction (Grade 2 or higher or per PI discretion) or anaphylaxis following administration of a vaccine.
* Severe asthma (defined as asthma that is unstable or required emergent care, urgent care, hospitalization, or intubation during the past two years, or that has required the use of oral or parenteral corticosteroids at any time during the past two years).
* Pre-existing autoimmune or antibody-mediated diseases including but not limited to:

systemic lupus erythematosus, rheumatoid arthritis, multiple sclerosis, Sjögren's syndrome, or autoimmune thrombocytopenia.

* Any confirmed or suspected immunosuppressive or immunodeficient state, including asplenia; recurrent, severe infections and chronic (more than 14 days) systemically active immunosuppressant medication within the past 6 months.
* Use of chronic (≥14 days) oral or IV corticosteroids (excluding topical or nasal) at immunosuppressive doses (i.e., prednisone ≥20 mg/day) or immunosuppressive drugs within 30 days of vaccination.
* Receipt of a live vaccine within the past 28 days or a killed vaccine within the past 14 days prior to Vaccination #1 and every subsequent vaccination day.
* Receipt of immunoglobulins and/or blood products within the past six months.
* Previous receipt of an investigational malaria vaccine in the last five years.
* Other condition(s) that, in the opinion of the investigator, would jeopardize the safety or rights of a participant participating in the trial, interfere with the evaluation of the study objectives, or would render the participant unable to comply with the protocol.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Healthy females of childbearing potential
Enrollment: 330 (Estimated)
Dates: Start 2025-03-19 (Actual); Primary Completion 2027-09-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of local and systemic solicited adverse events (AEs) | Within 7 days after each vaccine administration and over 6 months post third vaccination
  - Incidence of local and systemic solicited adverse events (AEs) graded by severity.
Number of participants with P falciparum infection | Over 6 months post third vaccination
  P. falciparum blood stage infection defined as time to first positive blood smear

SECONDARY OUTCOMES:
Assessment of safety and tolerabilty | Through study completion, an average of 26 months
  * Occurrence of unsolicited adverse events 28 days follow-up following the vaccination.
  * Occurrence of serious adverse events for the whole study duration including in women who become pregnant.
Anti-CSP antibody concentrations | Through study completion. Timepoints: baseline, days 70, 84, 140, 196, 434, 448, 504 and 560
  Immunological assessment measuring the anti-CSP antibody concentrations in healthy Malian women of child bearing potential
Rate of P.falciparum infection during pregnancy | Over 9-months pregnancy
  P. falciparum blood stage infection defined as time to first positive blood smear during pregnancy
Rate of P.falciparum infection | Over 12-, 18- and 24-months post third vaccination
  P. falciparum blood stage infection defined as time to first positive blood smear.

OTHER OUTCOMES:
Exploratory - number of participants with negative obstetric outcome | Over 9-months pregnancy
  negative maternal obstetric outcomes described as gestational diabetes, preterm premature rupture of membranes, third trimester hemorrhage, placental abruption, emergency C-section, post-partum hemorrhage, chorioamnionitis,miscarriage/stillbirth, intrauterine growth restriction, hypertensive diseases in pregnancy, preterm delivery
Exploratory - Immunology | Through study completion, an average of 26 months
  Antibody levels to VAR2CSA
Exploratory - Efficacy-Number of participants with symptomatic malaria | Through study completion, an average of 26 months
  - Symptomatic malaria defined as clinical or symptomatic malaria for this study is defined as the presence of asexual P. falciparum parasites at any parasitemia level and/or positive rapid diagnostic test with either an axillary temperature of 37.5 °C or more or one or more of the following symptoms: headache, myalgia, arthralgia, malaise, nausea, dizziness, or abdominal pain and will be reported as an AE
Exploratory - Efficacy-Number of participants with subclinical malaria infection | Through study completion, an average of 26 months
  P. falciparum qPCR may be performed from all scheduled visits with a malaria blood smear noted to capture infections that remain below the detection limit for microscopy
Exploratory - Efficacy-Number of participants with gametocytemia | Through study completion, an average of 26 months
  Blood smear microscopy to detect presence of P. falciparum gametocytes
Exploratory - Efficacy-Number of participants with non P. falciparum malaria infection | Through study completion, an average of 26 months
  Blood smear microscopy to detect presence of non-P. falciparum parasites
Exploratory - Efficacy-Number of infants with P falciparum infection | From birth until 12 months of age
  P. falciparum blood stage infection at blood smear during infancy
Exploratory - Efficacy-number of participants with P falciparum placental infection | Through study completion, an average of 26 months
  - P. falciparum placental infection defined as any positive placental blood smear for P. falciparum.
Exploratory - Number of babies with negative outcome | Up to 1 year
  negative neonatal outcome defined as neonatal death, low birth weight, small for gestational age, major malformations, hypoxic-ischemic encephalopathy, microcephaly, and APGAR score <7

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Hill, MD, Study Director — University of Oxford
Locations (1):
- Koumantou Study Clinic, Bougouni, Sikasso, Mali

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Datoo MS, Natama MH, Some A, Traore O, Rouamba T, Bellamy D, Yameogo P, Valia D, Tegneri M, Ouedraogo F, Soma R, Sawadogo S, Sorgho F, Derra K, Rouamba E, Orindi B, Ramos Lopez F, Flaxman A, Cappuccini F, Kailath R, Elias S, Mukhopadhyay E, Noe A, Cairns M, Lawrie A, Roberts R, Valea I, Sorgho H, Williams N, Glenn G, Fries L, Reimer J, Ewer KJ, Shaligram U, Hill AVS, Tinto H. Efficacy of a low-dose candidate malaria vaccine, R21 in adjuvant Matrix-M, with seasonal administration to children in Burkina Faso: a randomised controlled trial. Lancet. 2021 May 15;397(10287):1809-1818. doi: 10.1016/S0140-6736(21)00943-0. Epub 2021 May 5. PMID 33964223
- [Result] Datoo MS, Natama HM, Some A, Bellamy D, Traore O, Rouamba T, Tahita MC, Ido NFA, Yameogo P, Valia D, Millogo A, Ouedraogo F, Soma R, Sawadogo S, Sorgho F, Derra K, Rouamba E, Ramos-Lopez F, Cairns M, Provstgaard-Morys S, Aboagye J, Lawrie A, Roberts R, Valea I, Sorgho H, Williams N, Glenn G, Fries L, Reimer J, Ewer KJ, Shaligram U, Hill AVS, Tinto H. Efficacy and immunogenicity of R21/Matrix-M vaccine against clinical malaria after 2 years' follow-up in children in Burkina Faso: a phase 1/2b randomised controlled trial. Lancet Infect Dis. 2022 Dec;22(12):1728-1736. doi: 10.1016/S1473-3099(22)00442-X. Epub 2022 Sep 7. PMID 36087586